CLINICAL TRIAL: NCT04139824
Title: A Phase 1, Open-label, Fixed-sequence, 2-way Drug Interaction Study to Evaluate the Effect of Naproxen on the Pharmacokinetics of LC350189 and the Effect of LC350189 on the Pharmacokinetics of Naproxen in Healthy Subjects
Brief Title: The Effect of Naproxen on the Pharmacokinetic Profile of LC350189 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LG-GDCL006
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Anti-Inflammatory Agents, Non-Steroidal; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort (Experimental): Period 1: LC350189 200mg (QD) Day 1~ Day 4, Period 2: Naproxen 500 mg (BID) Day 8 ~ Day 12 , Period 3 : LC350189 200mg (QD) + Naproxen 500 mg (BID) Day 13~19
  Interventions: Drug: Xanthine Oxidase Inhibitor; Drug: nonsteroidal anti-inflammatory drug

INTERVENTIONS:
Drug: Xanthine Oxidase Inhibitor — LC350189 200mg qd
  Other Names: LC350189
Drug: nonsteroidal anti-inflammatory drug — Naproxen 500mg BID
  Other Names: Naproxen

SUMMARY:
This is a Phase 1, open-label, fixed-sequence, 3-period, 2-way drug interaction study designed to assess the pharmacokinetics, pharmacodynamics, safety, and tolerability of LC350189 and Naproxen when administered alone and in combination in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female 18 to 50 years of age, inclusive.
* The subject has a body mass index 18 to 32 kg/m2, inclusive, at screening.
* The subject is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12 lead electrocardiogram (ECG) results, and physical examination findings at screening.
* The subject agrees to comply with all protocol requirements.
* The subject is able to provide written informed consent.

Exclusion Criteria:

* The subject has a medical history with any issues affecting absorption or metabolism, as judged by the investigator.
* The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
* The subject has an estimated glomerular filtration rate (eGFR) of <90 (mL/min)/1.73 m2.
* The subject has used any prescription (excluding hormonal birth control and hormone replacement therapy) or over the counter medications (except paracetamol [up to 2 g per day]), including herbal or nutritional supplements, within 14 days before the first dose of study drug or throughout the study.
* The subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange containing products (eg, marmalade), or caffeine- or xanthine containing products within 48 hours before the first dose of study drug or throughout the study.
* The subject is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
* The subject has a history of alcohol abuse or drug addiction within the last year or excessive alcohol consumption (regular alcohol intake >21 units per week for male subjects and >14 units of alcohol per week for female subjects) (1 unit is equal to approximately ½ pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits).
* The subject has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at screening or before the first dose of study drug.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Maximun observed concentration (Cmax) of LC350189 and Naproxen from plasma | From baseline up to Day 18
  Pharmacokinetic
Area under the concentration-time curve (AUC) of LC350189 and Naproxen from plasma | From baseline up to Day 18
  Pharmacokinetic
Apparent terminal half-life (t1/2) of LC350189 and Naproxen from plasma | From baseline up to Day 18
  Pharmacokinetic

SECONDARY OUTCOMES:
Incidence of Adverse events | From baseline up to Day 18
  Safety
Changes in concentration of uric acid in plasma by uricase method | From baseline up to Day 17
  Pharmacodynamic

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided